CLINICAL TRIAL: NCT02531217
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, Biological Activity, and Systemic Exposure of ATYR1940 in Adult Patients With Fascioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Safety, Tolerability, Pharmacokinetics (PK), and Activity of ATYR1940 in Participants With Muscular Dystrophy - Study Extension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATYR1940-C-005; 2015-001912-36 (EudraCT Number)
Record Dates: First submitted 2015-06-25; First posted 2015-08-24 (Estimated); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATYR1940 (Experimental): Participants will receive ATYR1940 3.0 milligrams per kilograms (mg/kg) intravenous (IV) infusion once weekly for 24 weeks.
  Interventions: Biological: ATYR1940

INTERVENTIONS:
Biological: ATYR1940 — Concentrate for solution for infusion

SUMMARY:
The purpose of this study is to assess the safety and tolerability profile of ATYR1940 in the treatment of adult participants with molecularly defined genetic muscular dystrophies.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and tolerability profile of ATYR1940 in the treatment of adult participants with molecularly defined genetic muscular dystrophies, and to additionally explore the pharmacokinetics and biologic activity of ATYR1940 in adult participants with molecularly defined genetic muscular dystrophies. Participants who successfully complete the parent study (NCT02239224) are eligible for enrollment into this long-term extension study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has an established, genetically-confirmed, diagnosis of facioscapulohumeral dystrophy with clinical findings meeting existing criteria.
* Participant is a male or female aged 18 to 65 years, inclusive.
* Participants who previously participated in study ATYR1940-C-002 and who meet the entry criteria above for the current study will be eligible for enrollment.

Exclusion Criteria:

* Participant is currently receiving treatment with an immunomodulatory agent or has a history of such treatment, including targeted biological therapies (for example, etanercept, omalizumab) within the 3 months before Baseline; corticosteroids within 4 weeks before Baseline; or non-steroidal anti-inflammatory agents (NSAIDs) within 2 weeks before Baseline.
* Participant has a severe retinopathy.
* Participant has a history of obstructive or restrictive lung disease (including interstitial lung disease, pulmonary fibrosis, or asthma), or evidence for interstitial lung disease on Screening chest radiograph.
* Participant has evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, dermatological, or gastrointestinal disease, or has a condition that requires immediate surgical intervention, other treatment or may not allow safe participation.
* Participant has used any investigational product or device (other than a mobility assistance device) within 30 days before Baseline.
* If female and of childbearing potential (premenopausal and not surgically sterile), participant has a positive pregnancy test at Screening or is unwilling to use contraception from the time of Screening through the 1-month Follow-up visit. Acceptable methods of birth control include abstinence, barrier methods, hormones, or intra-uterine device.
* If male, participant is unwilling to use a condom plus spermicide during sexual intercourse from the time of Screening through the 1-month Follow-up visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- aTyr Pharma Investigative Site, Columbus, Ohio, United States
- aTyr Pharma Investigative Site, Rome, Italy
- aTyr Pharma Investigative Site, Nijmegen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who participated in Cohort 2 or 3, completed the double-blind treatment period and were considered to be compliant with the study drug by the Investigator in the Study ATYR1940-C-002 (NCT02239224) were eligible for participation in this study.
Groups:
- ATYR1940: Participants received ATYR1940 3.0 milligrams per kilograms (mg/kg) intravenous (IV) infusion once weekly for 24 weeks.
Period: Overall Study
Arm/Group | ATYR1940
Started | 9
Received at Least One Dose of Study Drug | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Groups:
- ATYR1940: Participants received ATYR1940 3.0 mg/kg IV infusion once weekly for 24 weeks.
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 53.2 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. AEs ware defined as any untoward medical occurrence in a participant administered study drug and that does not necessarily have a causal relationship with the study drug. Worsening of a pre-existing medical condition should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 36)
Population: ITT analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Participants
  TEAEs | 9
  SAEs | 0

2. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormality
Description: Body systems that were evaluated during the physical examination included general appearance, head, eyes, ears, nose, throat, cardiovascular system, respiratory system, gastrointestinal system (abdomen), lymphatic system, musculoskeletal system, skin, psychiatric, and neurologic. Neurologic examination included assessment of mental status, memory, cranial nerves, motor function, reflexes, and sensory testing. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Participants | 4

3. Primary Outcome: Number of Participants With a Vital Sign-Related Event Resulting in a TEAE
Description: The vital sign parameters that were evaluated included blood pressure, pulse and respiration rates, and body temperature. Vital signs abnormalities that were considered by the Investigator to be clinically significant were reported as AEs if the finding represented a change from baseline. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Participants | 0

4. Primary Outcome: Number of Participants With a Clinically Significant Pulmonary Function Event Resulting in a TEAE
Description: Pulmonary evaluations included pulmonary function tests. Clinically significant changes were to be reported as adverse events. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Participants | 0

5. Primary Outcome: Number of Participants With a Clinical Laboratory Abnormality Resulting in an AE
Description: Laboratory parameters included hematology (hematocrit, hemoglobin, red blood cell count, white blood cell count with differential [neutrophils, lymphocytes, monocytes, eosinophils, basophils], and platelet count); serum chemistries (blood urea nitrogen, creatinine, total bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, total protein, sodium, potassium, bicarbonate, calcium, chloride, magnesium, inorganic phosphate, creatine kinase, lactate dehydrogenase, C-reactive protein, troponin, myoglobin, insulin-like growth factor 1, and cholesterol [nonfasting]); and urinalysis (color, pH, specific gravity, protein, glucose, ketones, and blood). Clinically significant laboratory abnormalities were based upon Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 9
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to End of Study (up to Week 36)
Description: ITT analysis Set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Arm/Group | ATYR1940
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATYR1940 (N=9)
Ear Pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 2
Infusion Site Erythema (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 1
Ear Infection (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2
Muscle Injury (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Electrocardiogram QT Prolonged (Investigations) | 1
Hepatic Enzyme Increased (Investigations) | 2
Oxygen Saturation Decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 1
Muscle Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysstasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes